CLINICAL TRIAL: NCT04157348
Title: A Randomised, Double-blind, Active-controlled 52-week Study With an Open-label Extension to Evaluate the Efficacy and Safety of Benralizumab Compared to Mepolizumab in the Treatment of Eosinophilic Granulomatosis With Polyangiitis (EGPA) in Patients Receiving Standard of Care Therapy (MANDARA Study)
Brief Title: Efficacy and Safety of Benralizumab in EGPA Compared to Mepolizumab.
Acronym: MANDARA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3253C00001; 2023-510248-19-00 (Other: EU Trial (CTIS) Number); 2019-001832-77 (EudraCT Number)
Record Dates: First submitted 2019-09-29; First posted 2019-11-08 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Granulomatous Vasculitis
Keywords: Benralizumab; Inhaled corticosteroids; Eosinophilic Granulomatous Vasculitis
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — benralizumab; mepolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab arm (Experimental): 1x benralizumab SC injection + 3x placebo to mepolizumab SC injections
  Interventions: Biological: Benralizumab; Biological: Placebo to Mepolizumab
- Mepolizumab arm (Active Comparator): 3x mepolizumab SC injections + 1x placebo to benralizumab SC injection
  Interventions: Biological: Mepolizumab; Biological: Placebo to Benralizumab

INTERVENTIONS:
Biological: Benralizumab — 30 mg/mL solution for injection in a single accessorized prefilled syringe (APFS) will be administered subcutaneously (SC)
  Arms: Benralizumab arm
Biological: Mepolizumab — 3x100 mg vials of powder for solution for injection reconstituted into 3 separate 1 mL syringes for administration on each dosing occasion. Injection volume per syringe is 1 mL. Mepolizumab active solution will be administered subcutaneously (SC)
  Arms: Mepolizumab arm
Biological: Placebo to Mepolizumab — Matching placebo: 0.9% sodium chloride, solutions for injection in 1mL syringes (3 syringes will be used on each dosing occasion). Injection volume per syringe is 1mL. Placebo to Mepolizumban will be administered subcutaneously (SC)
  Arms: Benralizumab arm
Biological: Placebo to Benralizumab — Matching placebo solution for injection in APFS, 1 mL fill volume. Placebo solution will be administered subcutaneously (SC)
  Arms: Mepolizumab arm

SUMMARY:
This is a randomized, double blind, active-controlled, parallel group, multicenter 52-week Phase 3 study to compare the efficacy and safety of benralizumab 30 mg versus mepolizumab 300 mg administered by subcutaneous (SC) injection in patients with relapsing or refractory EGPA on corticosteroid therapy with or without stable immunosuppressive therapy.

All patients who complete the 52-week double-blind treatment period on IP may be eligible to continue into an open label extension (OLE) period. The OLE period is intended to allow each patient at least 1 year of treatment with open-label benralizumab 30 mg administered SC (earlier enrolled patients may therefore be in the OLE for longer than 1 year).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 18 years or older.
2. EGPA diagnosis based on history or presence asthma and eosinophilia (>1.0x10^9/L and/or >10% of leucocytes) and at least 2 of; biopsy with eosinophilic vasculitis or perivascular/granulomatous inflammation; mono-or polyneuropathy, non-fixed pulmonary infiltrates, sino-nasal abnormality; cardiomyopathy; glomerulonephritis; alveolar haemorrhage; palpable purpura; anti neutrophil cytoplasmic anti-body (ANCA) positivity (Myeloperoxidase or proteinease 3).
3. History of relapsing (at least 1 confirmed EGPA relapse within last 2 years and > 12 weeks prior to screening), or refractory (failure to attain remission, defined as BVAS=0 and oral corticosteroid (OCS) dose <=7.5 mg/day of prednisolone or equivalent, following standard induction regimen for at least 3 months and within 6 months prior to screening, or recurrence of symptoms upon OCS tapering at any dose of ≥7.5 mg/day prednisolone or equivalent.

   If induction with glucocorticoidsalone, patient must have failed to attain remission after 3 months and the glucocorticoid dose must be ≥15 mg/day prednisolone or equivalent for the 4 weeks prior to randomization.
4. Must be on a stable dose of oral prednisolone or prednisone of ≥7.5 mg/day (but not >50mg/day) for at least 4 weeks prior to randomization.
5. If receiving immunosuppressive therapy (excluding cyclophosphamide) the dose must be stable for the 4 weeks prior to randomization and during the study (dose reductions for safety reasons will be permitted).
6. QTc(F)<450 msec or QTc(F)<480 msec for patients with bundle branch block.
7. Females of childbearing potential must use an acceptable method of birth control from randomization for at least 12 weeks after the last study drug administration.

Exclusion Criteria:

1. Diagnosed with granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA)
2. Organ or life-threatening EGPA < 3 months prior to screening
3. Currently pregnant or breastfeeding, or planning to become pregnant during study participation.
4. Current malignancy or history of malignancy, unless received curative therapy >5 years ago, or >1 year ago for basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix
5. An untreated or refractory helminth parasitic infection < 24 weeks prior to screening
6. Unstable liver disease
7. Severe or clinically significant, uncontrolled cardiovascular disease
8. Other concurrent disease that may put the patient at risk, or may influence the results of the study, or the patients' ability to complete entire duration of the study
9. Chronic or ongoing infectious disease requiring systemic anti-infective treatment
10. Known immunodeficiency disorder or positive HIV test
11. Prior receipt of mepolizumab, reslizumab, dupilumab or benralizumab. Receipt of intravenous/intramuscular/subcutaneous corticosteroids within 4 weeks prior to randomization, receipt of omalizumab within 130 days prior to screening, rituximab within 6 months prior to screening (or B-cells not recovered), interferon-α or alemtuzumab within 6 months prior to screening, receipt of anti-tumor necrosis factor therapy within 12 weeks prior to screening or an investigational non-biologic product within 30 days or 5 half-lives prior to screening, whichever is longer. Receipt of any other marketed or investigational biologic products within 4 months or 5 half-lives prior to screening, whichever is longer.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wechsler, MD, Principal Investigator — National Jewish Health, 1400 Jackson St Denver, CO 80206
Locations (46):
- United States (9):
  - Research Site, Denver, Colorado
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Albuquerque, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Denison, Texas
  - Research Site, Seattle, Washington
- Research Site, Brussels, Belgium
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
- France (7):
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Suresnes
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Bamberg
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Kirchheim
  - Research Site, Lübeck
- Israel (6):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (6):
  - Research Site, Cuneo
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Torino
- Japan (5):
  - Research Site, Chiba
  - Research Site, Kita-gun
  - Research Site, Sagamihara-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Wechsler ME, Nair P, Terrier B, Walz B, Bourdin A, Jayne DRW, Jackson DJ, Roufosse F, Borjesson Sjo L, Fan Y, Jison M, McCrae C, Necander S, Shavit A, Walton C, Merkel PA; MANDARA Study Group. Benralizumab versus Mepolizumab for Eosinophilic Granulomatosis with Polyangiitis. N Engl J Med. 2024 Mar 7;390(10):911-921. doi: 10.1056/NEJMoa2311155. Epub 2024 Feb 23. PMID 38393328
- [Derived] Serling-Boyd N, Wallace ZS. Management of primary vasculitides with biologic and novel small molecule medications. Curr Opin Rheumatol. 2021 Jan;33(1):8-14. doi: 10.1097/BOR.0000000000000756. PMID 33164993
- See also: This is a poster. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3253C00001&attachmentIdentifier=f1ea6ab0-2192-44ba-9851-0549ffaf44a1&fileName=MANDARA_Poster_V2.0.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3253C00001&attachmentIdentifier=47896d32-8fa4-4f16-81e2-ded02ef2f949&fileName=d3253c00001-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 140 participants were randomized to receive treatment in study D3253C00001 (MANDARA) with benralizumab 30 mg or mepolizumab 300 mg. Of the 140 patients randomized, 140 (100%) received treatment with study drug. 70 (50%) patients received benralizumab 30 mg and 70 (50%) patients received mepolizumab 300 mg.
Pre-assignment Details: All patients completed a screening period of 1-4 weeks during which inclusion/exclusion criteria was assessed, disease activity, corticosteroid medication usage and patient reported outcomes were recorded, medical history and clinical laboratory were taken. All patients who entered open label extension period received benralizumab 30 mg during open label extension period.
Groups:
- Benralizumab 30 mg: Benralizumab and matching placebo injections delivered subcutaneously every 4 weeks
- Mepolizumab 300 mg: Mepolizumab and matching placebo injection delivered subcutaneously every 4 weeks
Period: Double-blind Treatment Period
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Started | 70 | 70
Completed | 69 | 67
Not Completed | 1 | 3
Not completed — other reasons or due to COVID-19 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Open-label Extension Period
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Started (Not all double-blind participants enrolled in the Open-label extension period) | 66 | 62
Completed (the study is still ongoing) | 0 | 0
Not Completed | 66 | 62
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Ongoing | 60 | 57
Not completed — other reasons | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received any IP were included in the full analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (13.90) | 52.7 (14.38) | 52.3 (14.10)
Age, Customized [Number; unit: participants]
  >= 18 to <= 65 years | 57 | 59 | 116
  > 65 years | 13 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 39 | 84
  Male | 25 | 31 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 61 | 67 | 128
  Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 53 | 57 | 110
  Asian | 9 | 8 | 17
  Other | 3 | 2 | 5
  Not reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  North America | 16 | 16 | 32
  Japan | 4 | 4 | 8
  Rest of World | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved Main Remission at Both Weeks 36 and 48
Description: Percentage of patients with relapsing or refractory EGPA, achieving remission, defined as BVAS = 0 and OCS dose ≤ 4 mg/day (main remission definition) at both Weeks 36 and 48.
Time Frame: Week 36 and Week 48
Population: Full Analysis Set: All patients randomized and receiving at least one (1) dose of IP are included in the full analysis set, irrespective of their protocol adherence and continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants | 40 | 40
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; Test type: Superiority; p = 0.8773, Regression, Logistic; marginal standardization method; Difference in remission rates = 0.0121, 95% CI 2-sided [-0.1411 to 0.1653] — The difference of remission rates (Benralizumab - Mepolizumab) are estimated using marginal standardization method in a logistic regression model. The covariates include treatment arm, baseline dose of prednisone, baseline BVAS and region

2. Primary Outcome: Supportive Endpoint: Proportion of Subjects Who Achieved Supportive Remission at Both Weeks 36 and 48
Description: Supportive endpoint: Proportion of patients with relapsing or refractory EGPA, achieving remission, defined as BVAS = 0 and OCS dose ≤ 7.5 mg/day (supportive remission definition) at both Weeks 36 and 48.
Time Frame: Week 36 and Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants | 55 | 52
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in remission rates = 0.0544, 95% CI 2-sided [-0.0746 to 0.1834]

3. Secondary Outcome: Total Accrued Duration of Remission During DB Treatment Period
Description: Total accrued duration of remission for the following categories: 0 week, > 0 to < 12 week, 12 to < 24 week, 24 to < 36 week, ≥ 36 week.
Time Frame: from baseline to end of DB period, 52 Weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  main remission: 0 week | 9 | 15
  main remission: >0 to <12 weeks | 13 | 10
  main remission: 12 to <24 weeks | 8 | 8
  main remission: 24 to <36 weeks | 20 | 19
  main remission: >=36 weeks | 20 | 18
  supportive remission: 0 week | 2 | 4
  supportive remission: >0 to <12 weeks | 2 | 3
  supportive remission: 12 to <24 weeks | 5 | 4
  supportive remission: 24 to <36 weeks | 16 | 15
  supportive remission: >=36 weeks | 45 | 44
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; main remission; Test type: Superiority; Proportional Odds Model; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.72 to 2.40] — The odds ratio (Benralizumab vs. Mepolizumab) and its 95% CI are estimated with a proportional odds model. The covariates include treatment arm, baseline dose of prednisone, baseline BVAS and region. A >1 odds ratio means Benralizumab is favored
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; supportive remission; Test type: Superiority; Proportional Odds Model; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.55 to 2.29] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Total Accrued Duration of Sustained Remission During DB Treatment Period
Description: Total accrued duration of sustained remission for the following categories: 0 week, > 0 to < 12 week, 12 to < 24 week, 24 to < 36 week, ≥ 36 week.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  sustained main remission: 0 week | 9 | 15
  sustained main remission: >0 to <12 weeks | 15 | 13
  sustained main remission: 12 to <24 weeks | 11 | 8
  sustained main remission: 24 to <36 weeks | 16 | 18
  sustained main remission: >=36 weeks | 19 | 16
  sustained supportive remission: 0 week | 2 | 4
  sustained supportive remission: >0 to <12 weeks | 5 | 6
  sustained supportive remission: 12 to <24 weeks | 8 | 10
  sustained supportive remission: 24 to <36 weeks | 18 | 14
  sustained supportive remission: >=36 weeks | 37 | 36
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; sustained main remission; Test type: Superiority; Proportional Odds Model; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.74 to 2.44] — The odds ratio (Benralizumab vs. Mepolizumab) and its 95% CI are estimated with a proportional odds model. The covariates include treatment arm, baseline dose of prednisone, baseline BVAS and region
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; sustained supportive remission; Test type: Superiority; Proportional Odds Model; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.64 to 2.34] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Time From Randomization to First Eosinophilic Granulomatosis With Polyangiitis (EGPA) Relapse
Description: Time from randomization to first Eosinophilic Granulomatosis with Polyangiitis (EGPA) relapse, where relapse is defined as any of the following:
  * Active vasculitis (BVAS > 0); OR
  * Active asthma symptoms and/or signs with a corresponding worsening in ACQ-6 score; OR
  * Active nasal and/or sinus disease, with a corresponding worsening in at least one of the sino-nasal symptom questions; warranting any of the following:
  * An increased dose of OCS therapy to > 4 mg/day prednisolone total daily dose; OR
  * An increased dose or addition of immunosuppressive therapy; OR
  * Hospitalization related to EGPA worsening Calculated using the Kaplan-Meier technique.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
percentage of subjects
  relapse-percent subject with at least 1 relapse by week 16 | 5.71 [2.18 to 14.51] | 4.29 [1.40 to 12.70]
  relapse-percent subject with at least 1 relapse by week 32 | 17.14 [10.12 to 28.21] | 20.24 [12.52 to 31.77]
  relapse-percent subject with at least 1 relapse by week 52 | 30.00 [20.71 to 42.21] | 29.10 [19.85 to 41.40]
  major relapse-percent subject with at least 1 relapse by week 16 | 0 [0 to 0] | 0 [0 to 0]
  major relapse-percent subject with at least 1 relapse by week 32 | 0 [0 to 0] | 0 [0 to 0]
  major relapse-percent subject with at least 1 relapse by week 52 | 0 [0 to 0] | 2.94 [0.74 to 11.25]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; relapse; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.53 to 1.82] — The HR (Benralizumab vs. Mepolizumab) and 95% CI are estimated using a Cox regression model with Efron method to control for ties. The covariates include treatment arm, baseline dose of prednisone, baseline BVAS and region

6. Secondary Outcome: Annualized Eosinophilic Granulomatosis With Polyangiitis (EGPA) Relapse Rate
Description: Annualized Eosinophilic Granulomatosis with Polyangiitis (EGPA) relapse rate through end of DB treatment period. The estimate of annualized relapse rate (relapses per year) and the corresponding 95% CIs were calculated using a negative binomial model. The response variable in the model is the number of relapses experienced by a subject up to Week 52. The logarithm of the subject's corresponding follow-up time up to Week 52 was used as an offset variable to adjust for subjects having different follow-up times during which the events occur. The covariates in the model include treatment arm, baseline dose of prednisone, baseline BVAS and region.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
relapses per year | 0.50 [0.30 to 0.83] | 0.49 [0.28 to 0.86]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; relapse; Test type: Superiority; negative binomial model; marginal standardization method; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.56 to 1.90] — The rate ratio (Benralizumab/Mepolizumab) and the corresponding 95% CI are calculated using a negative binomial model. The covariates in the model include treatment arm, baseline dose of prednisone, baseline BVAS and region

7. Secondary Outcome: Average Daily Dose of Prednisolone/Prednisone and Change From Baseline During Week 48 Through 52
Description: Average daily dose of prednisolone/prednisone and change from baseline during Week 48 through 52, or last 28 days prior to last double-blind assessment for those that withdrew
Time Frame: last 4 weeks of DB period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
mg
  average daily dose | 3.01 (3.776) | 3.43 (4.124)
  change from baseline of average daily dose | -8.08 (4.575) | -7.52 (7.070)

8. Secondary Outcome: Proportion of Patients With Average Daily Dose of Prednisolone/Prednisone During Week 48 Through 52
Description: Proportion of patients with average daily dose of prednisolone/prednisone during Week 48 through 52 in each category: 0 mg; >0 to ≤ 4 mg; > 4 to ≤ 7.5 mg and > 7.5 mg
Time Frame: last 4 weeks of DB period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  0 | 29 | 19
  >0 to <=4.0 mg | 19 | 30
  >4.0 to <=7.5 mg | 15 | 13
  >7.5 mg | 7 | 8
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; Test type: Superiority; proportional odds model; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.75 to 2.54] — The odds ratio (Benralizumab 30 mg vs. Mepolizumab 300 mg) and 95% CI are estimated using a proportional odds model. The covariates in the model include treatment arm, baseline dose of prednisone, baseline BVAS and region

9. Secondary Outcome: Percentage Reduction From Baseline in Average Daily Dose of Prednisolone/Prednisone During Week 48 Through 52
Description: Percentage reduction from baseline in average daily dose of prednisolone/prednisone during Week 48 through 52 in each category: no reduction or withdrawal from treatment; < 25% reduction; 25 to < 50% reduction; 50 to <75% reduction; 75 to < 100% reduction; 100% reduction.
Time Frame: last 4 weeks of DB period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  no reduction or withdrawal from IP before week 48 | 3 | 7
  <25% reduction | 0 | 2
  25 to <50% reduction | 8 | 9
  50 to <75% reduction | 19 | 17
  75 to <100% reduction | 11 | 17
  100% reduction | 29 | 18
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; Test type: Superiority; proportional odds model; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.96 to 3.22] — The odds ratio (Benralizumab 30 mg vs. Mepolizumab 300 mg) for higher % reduction and 95% CI are estimated using a proportional odds model. The covariates in the model include treatment arm, baseline dose of prednisone, baseline BVAS and region

10. Secondary Outcome: Proportion of Subjects With Reduction From Baseline in Average Daily Dose of Prednisolone/Prednisone During Week 48 Through 52
Description: Proportion of subjects with reduction from baseline in average daily dose of prednisolone/prednisone during Week 48 through 52 in each category: >= 50% reduction; 100% reduction; OCS dose <= 4 mg/day.
Time Frame: last 4 weeks of DB period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  >=50% reduction | 59 | 52
  100% reduction | 29 | 18
  OCS dose <=4 mg/day | 48 | 49
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; >=50% reduction; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in proportions = 0.1079, 95% CI 2-sided [-0.0225 to 0.2383] — The difference of proportions (Benralizumab - Mepolizumab) and 95% CI are estimated using marginal standardization method in a logistic regression model. The covariates include treatment arm, baseline dose of prednisone, baseline BVAS and region
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; 100% reduction; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in proportions = 0.1569, 95% CI 2-sided [0.0067 to 0.3017] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; OCS dose <=4 mg/day; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in proportions = -0.0068, 95% CI 2-sided [-0.1555 to 0.1418] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Proportion of Subjects Who Achieve Clinical Benefit
Description: Proportion of subjects who achieved any clinical benefit definition 1 (defined as any of the following:
  * Main remission at any time in DB period
  * >= 50% reduction in OCS dose in Weeks 48 to 52
  * EGPA relapse free in DB period) and subjects who achieved complete response definition 1 (defined as meeting all the definition 1 criteria above.)
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  any clinical benefit-definition 1 | 66 | 63
  Complete response - definition 1 | 43 | 39
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; any clinical response-definition 1; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in response rates = 0.046, 95% CI 2-sided [-0.0422 to 0.1341] — The difference of response rates (Benralizumab - Mepolizumab) and 95% CI are estimated using marginal standardization method in a logistic regression model. The covariates include treatment arm, baseline dose of prednisone, baseline BVAS and region
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; complete response-definition 1; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in response rates = 0.0790, 95% CI 2-sided [-0.0732 to 0.2312] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Proportion of Patients Who Have Achieved Remission Within the First 24 Weeks and Remained in Remission for Remainder of the Double-blind Treatment Period
Description: Proportion of patients who have achieved remission within the first 24 weeks and remained in remission for remainder of the double-blind treatment period
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  main remission | 28 | 27
  supportive remission | 41 | 40
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; main remission; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in remission rates = 0.0554, 95% CI 2-sided [-0.0930 to 0.2037] — The difference of remission rates (Benralizumab - Mepolizumab) and 95% CI are estimated using marginal standardization method in a logistic regression model. The covariates include treatment arm, baseline dose of prednisone, baseline BVAS and region
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Mepolizumab 300 mg; supportive remission; Test type: Superiority; Regression, Logistic; marginal standardization method; difference in remission rates = 0.0467, 95% CI 2-sided [-0.1021 to 0.1956] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Change From Baseline in Birmingham Vasculitis Activity Score (BVAS)
Description: Birmingham Vasculitis Activity Score (BVAS) change from baseline by timepoint up to week 52. The BVAS form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The total score on all 9 organ systems gives an indication of the disease activity of each patient at the time of scoring. Total scores range from 0 to 63, with higher scores indicating more active vasculitis.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
scores on a scale
  week 4 | -1.19 [-1.62 to -0.76] | -1.14 [-1.57 to -0.70]
  week 8 | -1.33 [-1.75 to -0.90] | -1.74 [-2.16 to -1.31]
  week 12 | -1.79 [-2.03 to -1.55] | -1.66 [-1.90 to -1.42]
  week 16 | -1.85 [-2.04 to -1.65] | -1.80 [-2.00 to -1.59]
  week 20 | -1.73 [-2.01 to -1.44] | -1.82 [-2.10 to -1.53]
  week 24 | -1.59 [-1.88 to -1.31] | -1.74 [-2.02 to -1.45]
  week 28 | -1.94 [-2.09 to -1.79] | -1.95 [-2.10 to -1.80]
  week 32 | -1.92 [-2.04 to -1.80] | -1.93 [-2.05 to -1.81]
  week 36 | -1.98 [-2.29 to -1.66] | -1.65 [-1.98 to -1.33]
  week 40 | -1.84 [-2.01 to -1.67] | -1.89 [-2.07 to -1.72]
  week 44 | -1.84 [-2.00 to -1.68] | -1.96 [-2.13 to -1.80]
  week 48 | -1.80 [-2.04 to -1.56] | -1.92 [-2.17 to -1.66]
  week 52 | -1.85 [-2.37 to -1.34] | -1.32 [-1.84 to -0.80]

14. Secondary Outcome: Spirometry Change From Baseline by Timepoint up to Week 52: Pre-BD FEV1 (L)
Description: Pre-bronchodilator (BD) Forced Expiratory Volume during first second (FEV1) change from baseline by timepoint up to week 52
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
L
  week 12 | 0.13 [0.0 to 0.2] | 0.11 [0.0 to 0.2]
  week 24 | 0.11 [0.0 to 0.2] | 0.13 [0.0 to 0.2]
  week 36 | 0.10 [-0.0 to 0.2] | 0.11 [0.0 to 0.2]
  week 48 | 0.03 [-0.1 to 0.1] | 0.06 [-0.0 to 0.2]
  week 52 | 0.06 [-0.0 to 0.2] | 0.01 [-0.1 to 0.1]

15. Secondary Outcome: Spirometry Change From Baseline by Timepoint up to Week 52: Pre-BD FVC (L)
Description: Pre-bronchodilator (BD) Forced vital capacity (FVC) change from baseline by timepoint up to week 52
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
L
  week 12 | 0.13 [0.0 to 0.2] | 0.05 [-0.0 to 0.2]
  week 24 | 0.09 [0.0 to 0.2] | 0.04 [-0.1 to 0.1]
  week 36 | 0.05 [-0.0 to 0.1] | 0.03 [-0.1 to 0.1]
  week 48 | 0.03 [-0.1 to 0.1] | 0.00 [-0.1 to 0.1]
  week 52 | 0.01 [-0.1 to 0.1] | -0.04 [-0.2 to 0.1]

16. Secondary Outcome: Change From Baseline in Vasculitis Damage Index (VDI)
Description: Vasculitis Damage Index (VDI) change from baseline by timepoint up to week 52. The VDI is divided into 11 organ systems and records items of damage, due to vasculitis, treatment or unrelated, that have occurred since the onset of vasculitis. Completion of the form provides a numerical score, ranging from 0 to 64, with a higher score indicating more damage.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 24 | 0.06 [-0.00 to 0.12] | 0.04 [-0.02 to 0.10]
  week 52 | 0.13 [0.04 to 0.22] | 0.10 [0.01 to 0.20]

17. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (6-item Version) (ACQ-6)
Description: Asthma Control Questionnaire (6-item version) (ACQ-6) change from baseline by timepoint up to week 52. The ACQ-6 score is calculated by taking the mean of 6 equally weighted domains, with a range of 0 (well controlled) to 6 (extremely poorly controlled).
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 1-4 | -0.34 [-0.47 to -0.21] | -0.31 [-0.44 to -0.18]
  week 5-8 | -0.56 [-0.68 to -0.43] | -0.49 [-0.61 to -0.36]
  week 9-12 | -0.55 [-0.68 to -0.42] | -0.52 [-0.65 to -0.39]
  week 13-16 | -0.62 [-0.76 to -0.48] | -0.48 [-0.62 to -0.33]
  week 17-20 | -0.59 [-0.75 to -0.43] | -0.47 [-0.63 to -0.31]
  week 21-24 | -0.59 [-0.76 to -0.43] | -0.53 [-0.70 to -0.37]
  week 25-28 | -0.65 [-0.80 to -0.49] | -0.49 [-0.64 to -0.33]
  week 29-32 | -0.56 [-0.73 to -0.39] | -0.50 [-0.67 to -0.33]
  week 33-36 | -0.57 [-0.73 to -0.41] | -0.55 [-0.71 to -0.39]
  week 37-40 | -0.57 [-0.72 to -0.42] | -0.54 [-0.69 to -0.39]
  week 41-44 | -0.58 [-0.73 to -0.43] | -0.60 [-0.75 to -0.45]
  week 45-48 | -0.61 [-0.76 to -0.45] | -0.64 [-0.79 to -0.48]
  week 49-52 | -0.57 [-0.72 to -0.41] | -0.61 [-0.77 to -0.46]

18. Secondary Outcome: Change From Baseline in Short Form 36-item Health Survey (Version 2, Acute Recall) (SF-36v2) Component: Physical Component Summary (PCS)
Description: Short Form 36-item health survey (version 2, acute recall) (SF-36v2) component Physical Component Summary (PCS) change from baseline by timepoint up to week 52. PCS score ranges from 10.8 to 75.5, where a higher score indicates better health.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 1 | 0.68 [-0.4 to 1.7] | 0.88 [-0.2 to 1.9]
  week 4 | 1.18 [-0.1 to 2.5] | 1.11 [-0.2 to 2.4]
  week 8 | 1.56 [0.3 to 2.8] | 1.46 [0.2 to 2.7]
  week 12 | 1.30 [-0.0 to 2.6] | 1.31 [-0.0 to 2.6]
  week 16 | 1.24 [-0.2 to 2.7] | 1.85 [0.4 to 3.3]
  week 28 | 1.54 [-0.0 to 3.1] | 2.12 [0.6 to 3.7]
  week 40 | 1.73 [0.4 to 3.1] | 2.28 [0.9 to 3.6]
  week 52 | 0.29 [-1.3 to 1.9] | 2.45 [0.8 to 4.0]

19. Secondary Outcome: Change From Baseline in Short Form 36-item Health Survey (Version 2, Acute Recall) (SF-36v2) Component: Mental Component Summary (MCS)
Description: Short Form 36-item health survey (version 2, acute recall) (SF-36v2) component Mental Component Summary (MCS) change from baseline by timepoint up to week 52. MCS score ranges from 5.6 to 69.7, where a higher score indicates better health.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 1 | 0.90 [-0.7 to 2.5] | -0.13 [-1.7 to 1.5]
  week 4 | 0.06 [-1.8 to 1.9] | 0.58 [-1.2 to 2.4]
  week 8 | 0.64 [-1.3 to 2.6] | 1.05 [-0.9 to 3.0]
  week 12 | 0.04 [-1.9 to 2.0] | 1.44 [-0.5 to 3.4]
  week 16 | 0.29 [-1.8 to 2.3] | 2.18 [0.1 to 4.2]
  week 28 | -0.03 [-2.0 to 1.9] | 2.03 [0.1 to 4.0]
  week 40 | 0.77 [-1.5 to 3.0] | 2.39 [0.2 to 4.6]
  week 52 | 1.13 [-1.1 to 3.4] | 2.19 [-0.1 to 4.4]

20. Secondary Outcome: Change From Baseline in Sino-nasal Outcome Test-22 (SNOT-22) Total Score
Description: Sino-nasal Outcome Test-22 (SNOT-22) total score change from baseline by timepoint up to week 52. Patient reported symptom severity and symptom impact over the previous 2 weeks on 22 items are captured via a 6-point scale (0 = no problem to 5 = problem as bad as it can be). The total score is the sum of item scores and ranges from 0 to 110 (higher scores indicate poorer outcomes).
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 4 | -4.34 [-7.2 to -1.5] | -4.32 [-7.2 to -1.5]
  week 8 | -5.79 [-8.8 to -2.8] | -6.42 [-9.4 to -3.4]
  week 12 | -5.30 [-8.5 to -2.1] | -6.35 [-9.5 to -3.2]
  week 16 | -6.04 [-9.2 to -2.9] | -6.04 [-9.2 to -2.9]
  week 28 | -7.89 [-11.0 to -4.8] | -7.59 [-10.7 to -4.5]
  week 40 | -5.05 [-8.2 to -1.9] | -8.33 [-11.6 to -5.1]
  week 52 | -5.98 [-9.3 to -2.7] | -6.35 [-9.7 to -3.0]

21. Secondary Outcome: Sino-nasal Symptoms Questionnaire (SSQ) Scores: Symptom Runny Nose
Description: Sino-nasal Symptoms Questionnaire (SSQ) scores : symptom runny nose by timepoint. For the SSQ, participants rate each symptom against the following categories: very severe, severe, moderate, mild, none. Higher scores indicate greater severity (0 = none to 4 = very severe).
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  baseline | 1.0 (0.85) | 1.2 (1.00)
  week 1-4 | 1.4 (0.95) | 1.2 (0.97)
  week 5-8 | 1.3 (0.92) | 1.0 (0.86)
  week 9-12 | 1.4 (1.00) | 1.0 (0.88)
  week 13-16 | 1.4 (0.99) | 1.2 (0.92)
  week 17-20 | 1.3 (0.98) | 1.1 (0.96)
  week 21-24 | 1.3 (0.88) | 1.2 (0.86)
  week 25-28 | 1.1 (0.95) | 1.2 (0.90)
  week 29-32 | 1.2 (0.90) | 1.1 (0.99)
  week 33-36 | 1.3 (0.87) | 1.0 (0.90)
  week 37-40 | 1.3 (0.96) | 1.0 (0.87)
  week 41-44 | 1.1 (0.86) | 0.9 (0.76)
  week 45-48 | 1.3 (0.98) | 0.9 (0.87)
  week 49-52 | 1.2 (0.98) | 1.0 (0.96)

22. Secondary Outcome: Sino-nasal Symptoms Questionnaire (SSQ) Scores: Symptom Post-nasal Discharge
Description: Sino-nasal Symptoms Questionnaire (SSQ) scores : symptom Post-nasal discharge by timepoint. For the SSQ, participants rate each symptom against the following categories: very severe, severe, moderate, mild, none. Higher scores indicate greater severity (0 = none to 4 = very severe).
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  baseline | 1.1 (1.00) | 1.2 (1.06)
  week 1-4 | 1.4 (0.88) | 1.3 (1.00)
  week 5-8 | 1.2 (0.94) | 1.2 (0.85)
  week 9-12 | 1.2 (1.01) | 1.2 (0.98)
  week 13-16 | 1.2 (0.96) | 1.2 (0.94)
  week 17-20 | 1.2 (0.99) | 1.3 (0.99)
  week 21-24 | 1.2 (0.93) | 1.2 (0.98)
  week 25-28 | 1.1 (1.05) | 1.1 (0.88)
  week 29-32 | 1.1 (0.97) | 1.1 (0.99)
  week 33-36 | 1.1 (0.88) | 1.0 (0.95)
  week 37-40 | 1.2 (0.96) | 0.9 (0.81)
  week 41-44 | 1.1 (1.05) | 0.9 (0.83)
  week 45-48 | 1.1 (1.03) | 1.0 (0.89)
  week 49-52 | 1.1 (0.96) | 1.0 (0.95)

23. Secondary Outcome: Sino-nasal Symptoms Questionnaire (SSQ) Scores: Symptom Facial Pain/Pressure
Description: Sino-nasal Symptoms Questionnaire (SSQ) scores: symptom Facial pain/pressure by timepoint. For the SSQ, participants rate each symptom against the following categories: very severe, severe, moderate, mild, none. Higher scores indicate greater severity (0 = none to 4 = very severe).
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  baseline | 0.7 (0.95) | 0.6 (0.94)
  week 1-4 | 0.9 (0.97) | 0.8 (0.99)
  week 5-8 | 0.9 (1.08) | 0.8 (0.93)
  week 9-12 | 0.9 (1.01) | 0.8 (0.88)
  week 13-16 | 0.8 (0.93) | 0.6 (0.80)
  week 17-20 | 0.9 (0.97) | 0.7 (0.93)
  week 21-24 | 0.8 (0.88) | 0.6 (0.81)
  week 25-28 | 0.7 (0.95) | 0.6 (0.89)
  week 29-32 | 0.7 (0.89) | 0.6 (0.90)
  week 33-36 | 0.6 (0.86) | 0.6 (0.89)
  week 37-40 | 0.8 (1.01) | 0.6 (0.82)
  week 41-44 | 0.7 (0.92) | 0.6 (0.82)
  week 45-48 | 0.7 (0.90) | 0.7 (0.98)
  week 49-52 | 0.7 (0.90) | 0.6 (0.87)

24. Secondary Outcome: Sino-nasal Symptoms Questionnaire (SSQ) Scores: Symptom Loss or Reduction in Sense of Taste/Smell
Description: Sino-nasal Symptoms Questionnaire (SSQ) scores: symptom Loss or reduction in sense of taste/smell by timepoint. For the SSQ, participants rate each symptom against the following categories: very severe, severe, moderate, mild, none. Higher scores indicate greater severity (0 = none to 4 = very severe).
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  baseline | 1.3 (1.32) | 1.2 (1.43)
  week 1-4 | 1.3 (1.36) | 1.2 (1.45)
  week 5-8 | 1.2 (1.28) | 1.1 (1.35)
  week 9-12 | 1.2 (1.29) | 1.0 (1.36)
  week 13-16 | 1.3 (1.32) | 1.1 (1.41)
  week 17-20 | 1.3 (1.36) | 1.1 (1.32)
  week 21-24 | 1.4 (1.44) | 1.2 (1.33)
  week 25-28 | 1.3 (1.39) | 1.1 (1.37)
  week 29-32 | 1.4 (1.34) | 1.0 (1.38)
  week 33-36 | 1.4 (1.39) | 1.1 (1.35)
  week 37-40 | 1.5 (1.38) | 1.1 (1.31)
  week 41-44 | 1.5 (1.43) | 1.0 (1.29)
  week 45-48 | 1.5 (1.44) | 1.1 (1.36)
  week 49-52 | 1.5 (1.40) | 1.1 (1.35)

25. Secondary Outcome: Sino-nasal Symptoms Questionnaire (SSQ) Scores: Symptom Blockage/Congestion of Nose
Description: Sino-nasal Symptoms Questionnaire (SSQ) scores: symptom Blockage/congestion of nose by timepoint. For the SSQ, participants rate each symptom against the following categories: very severe, severe, moderate, mild, none. Higher scores indicate greater severity (0 = none to 4 = very severe).
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  baseline | 1.3 (1.07) | 1.4 (1.15)
  week 1-4 | 1.5 (0.99) | 1.4 (0.96)
  week 5-8 | 1.5 (0.96) | 1.4 (1.03)
  week 9-12 | 1.5 (0.90) | 1.3 (1.00)
  week 13-16 | 1.6 (1.14) | 1.4 (1.09)
  week 17-20 | 1.7 (1.12) | 1.4 (1.04)
  week 21-24 | 1.6 (1.06) | 1.3 (1.05)
  week 25-28 | 1.4 (1.03) | 1.4 (1.03)
  week 29-32 | 1.5 (0.99) | 1.4 (1.13)
  week 33-36 | 1.5 (0.92) | 1.3 (1.09)
  week 37-40 | 1.6 (1.01) | 1.3 (1.14)
  week 41-44 | 1.5 (1.08) | 1.2 (0.96)
  week 45-48 | 1.5 (1.13) | 1.3 (1.11)
  week 49-52 | 1.5 (1.07) | 1.3 (1.03)

26. Secondary Outcome: Patient Global Impression of Severity (PGIS) Category
Description: Patient Global Impression of Severity (PGIS) category by timepoint
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  baseline: No symptoms | 8 | 2
  baseline: Very mild | 8 | 19
  baseline: Mild | 18 | 16
  baseline: Moderate | 28 | 26
  baseline: Severe | 7 | 5
  baseline: Very severe | 1 | 2
  baseline: Missing | 0 | 0
  week 1: No symptoms | 4 | 4
  week 1: Very mild | 15 | 15
  week 1: Mild | 21 | 16
  week 1: Moderate | 24 | 26
  week 1: Severe | 4 | 6
  week 1: Very severe | 1 | 0
  week 1: Missing | 1 | 3
  week 2: No symptoms | 12 | 5
  week 2: Very mild | 14 | 27
  week 2: Mild | 21 | 11
  week 2: Moderate | 20 | 18
  week 2: Severe | 1 | 3
  week 2: Very severe | 0 | 1
  week 2: Missing | 2 | 5
  week 3: No symptoms | 9 | 8
  week 3: Very mild | 23 | 24
  week 3: Mild | 16 | 19
  week 3: Moderate | 18 | 13
  week 3: Severe | 2 | 3
  week 3: Very severe | 0 | 0
  week 3: Missing | 2 | 3
  week 4: No symptoms | 6 | 8
  week 4: Very mild | 17 | 20
  week 4: Mild | 15 | 13
  week 4: Moderate | 26 | 23
  week 4: Severe | 3 | 5
  week 4: Very severe | 1 | 0
  week 4: Missing | 2 | 1
  week 5: No symptoms | 12 | 6
  week 5: Very mild | 20 | 31
  week 5: Mild | 24 | 15
  week 5: Moderate | 12 | 14
  week 5: Severe | 0 | 3
  week 5: Very severe | 0 | 0
  week 5: Missing | 2 | 1
  week 6: No symptoms | 8 | 9
  week 6: Very mild | 29 | 33
  week 6: Mild | 18 | 13
  week 6: Moderate | 13 | 9
  week 6: Severe | 1 | 1
  week 6: Very severe | 0 | 2
  week 6: Missing | 1 | 3
  week 7: No symptoms | 8 | 12
  week 7: Very mild | 25 | 23
  week 7: Mild | 18 | 20
  week 7: Moderate | 14 | 10
  week 7: Severe | 3 | 1
  week 7: Very severe | 0 | 1
  week 7: Missing | 2 | 3
  week 8: No symptoms | 4 | 5
  week 8: Very mild | 18 | 24
  week 8: Mild | 18 | 15
  week 8: Moderate | 21 | 20
  week 8: Severe | 6 | 3
  week 8: Very severe | 1 | 2
  week 8: Missing | 2 | 1
  week 9: No symptoms | 7 | 14
  week 9: Very mild | 26 | 22
  week 9: Mild | 17 | 17
  week 9: Moderate | 14 | 13
  week 9: Severe | 4 | 2
  week 9: Very severe | 0 | 0
  week 9: Missing | 2 | 2
  week 10: No symptoms | 7 | 11
  week 10: Very mild | 21 | 24
  week 10: Mild | 24 | 22
  week 10: Moderate | 13 | 7
  week 10: Severe | 1 | 2
  week 10: Very severe | 2 | 0
  week 10: Missing | 2 | 4
  week 11: No symptoms | 7 | 13
  week 11: Very mild | 27 | 24
  week 11: Mild | 17 | 15
  week 11: Moderate | 14 | 15
  week 11: Severe | 2 | 1
  week 11: Very severe | 1 | 0
  week 11: Missing | 2 | 2
  week 12: No symptoms | 6 | 8
  week 12: Very mild | 18 | 20
  week 12: Mild | 19 | 16
  week 12: Moderate | 17 | 20
  week 12: Severe | 6 | 4
  week 12: Very severe | 2 | 0
  week 12: Missing | 2 | 2
  week 13: No symptoms | 6 | 9
  week 13: Very mild | 26 | 24
  week 13: Mild | 22 | 18
  week 13: Moderate | 11 | 15
  week 13: Severe | 2 | 3
  week 13: Very severe | 1 | 0
  week 13: Missing | 2 | 1
  week 14: No symptoms | 6 | 11
  week 14: Very mild | 29 | 24
  week 14: Mild | 15 | 15
  week 14: Moderate | 15 | 15
  week 14: Severe | 2 | 1
  week 14: Very severe | 0 | 1
  week 14: Missing | 3 | 3
  week 15: No symptoms | 6 | 11
  week 15: Very mild | 31 | 23
  week 15: Mild | 12 | 17
  week 15: Moderate | 16 | 16
  week 15: Severe | 3 | 1
  week 15: Very severe | 0 | 0
  week 15: Missing | 2 | 2
  week 16: No symptoms | 3 | 5
  week 16: Very mild | 23 | 21
  week 16: Mild | 17 | 26
  week 16: Moderate | 19 | 13
  week 16: Severe | 5 | 1
  week 16: Very severe | 1 | 1
  week 16: Missing | 2 | 3
  week 17: No symptoms | 13 | 6
  week 17: Very mild | 23 | 28
  week 17: Mild | 14 | 19
  week 17: Moderate | 19 | 11
  week 17: Severe | 1 | 2
  week 17: Very severe | 0 | 1
  week 17: Missing | 0 | 3
  week 18: No symptoms | 7 | 7
  week 18: Very mild | 27 | 28
  week 18: Mild | 14 | 13
  week 18: Moderate | 18 | 18
  week 18: Severe | 0 | 2
  week 18: Very severe | 2 | 0
  week 18: Missing | 2 | 2
  week 19: No symptoms | 7 | 11
  week 19: Very mild | 27 | 25
  week 19: Mild | 14 | 17
  week 19: Moderate | 14 | 15
  week 19: Severe | 5 | 0
  week 19: Very severe | 2 | 1
  week 19: Missing | 1 | 1
  week 20: No symptoms | 8 | 13
  week 20: Very mild | 22 | 20
  week 20: Mild | 18 | 21
  week 20: Moderate | 14 | 11
  week 20: Severe | 7 | 1
  week 20: Very severe | 0 | 1
  week 20: Missing | 1 | 3
  week 21: No symptoms | 7 | 15
  week 21: Very mild | 26 | 24
  week 21: Mild | 13 | 12
  week 21: Moderate | 17 | 13
  week 21: Severe | 5 | 2
  week 21: Very severe | 1 | 0
  week 21: Missing | 1 | 4
  week 22: No symptoms | 13 | 12
  week 22: Very mild | 19 | 24
  week 22: Mild | 19 | 16
  week 22: Moderate | 16 | 12
  week 22: Severe | 3 | 1
  week 22: Very severe | 0 | 0
  week 22: Missing | 0 | 5
  week 23: No symptoms | 8 | 13
  week 23: Very mild | 24 | 24
  week 23: Mild | 20 | 19
  week 23: Moderate | 14 | 13
  week 23: Severe | 1 | 1
  week 23: Very severe | 2 | 0
  week 23: Missing | 1 | 0
  week 24: No symptoms | 7 | 13
  week 24: Very mild | 25 | 22
  week 24: Mild | 20 | 16
  week 24: Moderate | 14 | 16
  week 24: Severe | 3 | 2
  week 24: Very severe | 0 | 0
  week 24: Missing | 1 | 1
  week 25: No symptoms | 11 | 13
  week 25: Very mild | 25 | 22
  week 25: Mild | 19 | 17
  week 25: Moderate | 10 | 14
  week 25: Severe | 4 | 0
  week 25: Very severe | 0 | 0
  week 25: Missing | 1 | 4
  week 26: No symptoms | 12 | 13
  week 26: Very mild | 25 | 22
  week 26: Mild | 17 | 14
  week 26: Moderate | 11 | 15
  week 26: Severe | 3 | 2
  week 26: Very severe | 1 | 1
  week 26: Missing | 1 | 3
  week 27: No symptoms | 10 | 15
  week 27: Very mild | 28 | 21
  week 27: Mild | 16 | 17
  week 27: Moderate | 15 | 10
  week 27: Severe | 0 | 2
  week 27: Very severe | 1 | 0
  week 27: Missing | 0 | 5
  week 28: No symptoms | 6 | 9
  week 28: Very mild | 21 | 21
  week 28: Mild | 23 | 18
  week 28: Moderate | 14 | 16
  week 28: Severe | 4 | 2
  week 28: Very severe | 1 | 0
  week 28: Missing | 1 | 4
  week 29: No symptoms | 6 | 12
  week 29: Very mild | 28 | 21
  week 29: Mild | 17 | 19
  week 29: Moderate | 15 | 10
  week 29: Severe | 2 | 3
  week 29: Very severe | 0 | 0
  week 29: Missing | 2 | 5
  week 30: No symptoms | 7 | 18
  week 30: Very mild | 22 | 16
  week 30: Mild | 25 | 18
  week 30: Moderate | 11 | 9
  week 30: Severe | 3 | 2
  week 30: Very severe | 0 | 1
  week 30: Missing | 2 | 6
  week 31: No symptoms | 8 | 16
  week 31: Very mild | 22 | 20
  week 31: Mild | 18 | 17
  week 31: Moderate | 16 | 11
  week 31: Severe | 3 | 2
  week 31: Very severe | 0 | 0
  week 31: Missing | 3 | 4
  week 32: No symptoms | 6 | 15
  week 32: Very mild | 25 | 20
  week 32: Mild | 17 | 20
  week 32: Moderate | 16 | 8
  week 32: Severe | 3 | 3
  week 32: Very severe | 1 | 0
  week 32: Missing | 2 | 4
  week 33: No symptoms | 6 | 17
  week 33: Very mild | 23 | 20
  week 33: Mild | 22 | 14
  week 33: Moderate | 14 | 13
  week 33: Severe | 2 | 1
  week 33: Very severe | 0 | 0
  week 33: Missing | 3 | 5
  week 34: No symptoms | 8 | 14
  week 34: Very mild | 27 | 18
  week 34: Mild | 17 | 20
  week 34: Moderate | 13 | 11
  week 34: Severe | 2 | 2
  week 34: Very severe | 1 | 0
  week 34: Missing | 2 | 5
  week 35: No symptoms | 10 | 16
  week 35: Very mild | 25 | 20
  week 35: Mild | 16 | 18
  week 35: Moderate | 13 | 10
  week 35: Severe | 2 | 2
  week 35: Very severe | 1 | 0
  week 35: Missing | 3 | 4
  week 36: No symptoms | 7 | 15
  week 36: Very mild | 26 | 22
  week 36: Mild | 15 | 17
  week 36: Moderate | 18 | 12
  week 36: Severe | 1 | 1
  week 36: Very severe | 1 | 0
  week 36: Missing | 2 | 3
  week 37: No symptoms | 5 | 17
  week 37: Very mild | 28 | 21
  week 37: Mild | 18 | 14
  week 37: Moderate | 15 | 11
  week 37: Severe | 1 | 2
  week 37: Very severe | 0 | 1
  week 37: Missing | 3 | 4
  week 38: No symptoms | 7 | 17
  week 38: Very mild | 25 | 24
  week 38: Mild | 16 | 10
  week 38: Moderate | 16 | 12
  week 38: Severe | 1 | 3
  week 38: Very severe | 0 | 0
  week 38: Missing | 5 | 4
  week 39: No symptoms | 5 | 19
  week 39: Very mild | 30 | 23
  week 39: Mild | 14 | 13
  week 39: Moderate | 16 | 9
  week 39: Severe | 1 | 2
  week 39: Very severe | 0 | 0
  week 39: Missing | 4 | 4
  week 40: No symptoms | 2 | 10
  week 40: Very mild | 20 | 18
  week 40: Mild | 24 | 18
  week 40: Moderate | 18 | 14
  week 40: Severe | 2 | 3
  week 40: Very severe | 0 | 1
  week 40: Missing | 4 | 6
  week 41: No symptoms | 6 | 17
  week 41: Very mild | 25 | 23
  week 41: Mild | 20 | 16
  week 41: Moderate | 13 | 4
  week 41: Severe | 1 | 5
  week 41: Very severe | 0 | 0
  week 41: Missing | 5 | 5
  week 42: No symptoms | 7 | 15
  week 42: Very mild | 23 | 26
  week 42: Mild | 18 | 17
  week 42: Moderate | 15 | 4
  week 42: Severe | 2 | 3
  week 42: Very severe | 0 | 0
  week 42: Missing | 5 | 5
  week 43: No symptoms | 9 | 15
  week 43: Very mild | 17 | 27
  week 43: Mild | 21 | 16
  week 43: Moderate | 13 | 6
  week 43: Severe | 1 | 2
  week 43: Very severe | 2 | 0
  week 43: Missing | 7 | 4
  week 44: No symptoms | 6 | 16
  week 44: Very mild | 24 | 23
  week 44: Mild | 19 | 17
  week 44: Moderate | 14 | 6
  week 44: Severe | 2 | 3
  week 44: Very severe | 1 | 0
  week 44: Missing | 4 | 5
  week 45: No symptoms | 8 | 16
  week 45: Very mild | 21 | 26
  week 45: Mild | 22 | 14
  week 45: Moderate | 13 | 8
  week 45: Severe | 2 | 3
  week 45: Very severe | 0 | 0
  week 45: Missing | 4 | 3
  week 46: No symptoms | 9 | 16
  week 46: Very mild | 23 | 27
  week 46: Mild | 13 | 15
  week 46: Moderate | 17 | 7
  week 46: Severe | 3 | 2
  week 46: Very severe | 1 | 0
  week 46: Missing | 4 | 3
  week 47: No symptoms | 6 | 17
  week 47: Very mild | 25 | 27
  week 47: Mild | 16 | 11
  week 47: Moderate | 16 | 7
  week 47: Severe | 2 | 2
  week 47: Very severe | 1 | 0
  week 47: Missing | 4 | 6
  week 48: No symptoms | 11 | 17
  week 48: Very mild | 26 | 23
  week 48: Mild | 14 | 13
  week 48: Moderate | 15 | 9
  week 48: Severe | 1 | 4
  week 48: Very severe | 2 | 0
  week 48: Missing | 1 | 4
  week 49: No symptoms | 12 | 14
  week 49: Very mild | 20 | 25
  week 49: Mild | 18 | 16
  week 49: Moderate | 15 | 10
  week 49: Severe | 2 | 0
  week 49: Very severe | 0 | 0
  week 49: Missing | 3 | 5
  week 50: No symptoms | 10 | 16
  week 50: Very mild | 29 | 26
  week 50: Mild | 12 | 13
  week 50: Moderate | 15 | 8
  week 50: Severe | 1 | 0
  week 50: Very severe | 1 | 1
  week 50: Missing | 2 | 6
  week 51: No symptoms | 12 | 15
  week 51: Very mild | 18 | 25
  week 51: Mild | 16 | 16
  week 51: Moderate | 16 | 3
  week 51: Severe | 2 | 2
  week 51: Very severe | 0 | 0
  week 51: Missing | 6 | 9
  week 52: No symptoms | 4 | 11
  week 52: Very mild | 20 | 18
  week 52: Mild | 14 | 19
  week 52: Moderate | 16 | 12
  week 52: Severe | 5 | 1
  week 52: Very severe | 2 | 0
  week 52: Missing | 9 | 9

27. Secondary Outcome: Patient Global Impression of Change (PGIC) Category
Description: Patient Global Impression of Change (PGIC) category by timepoint
Time Frame: from baseline to week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
Participants
  week 1: Much better | 2 | 0
  week 1: Moderately better | 4 | 1
  week 1: A little better | 15 | 21
  week 1: About the same | 45 | 39
  week 1: A little worse | 2 | 5
  week 1: Moderately worse | 1 | 0
  week 1: Much worse | 0 | 0
  week 1: Missing | 1 | 4
  week 2: Much better | 7 | 2
  week 2: Moderately better | 7 | 6
  week 2: A little better | 14 | 22
  week 2: About the same | 38 | 33
  week 2: A little worse | 2 | 1
  week 2: Moderately worse | 0 | 0
  week 2: Much worse | 0 | 1
  week 2: Missing | 2 | 5
  week 3: Much better | 7 | 3
  week 3: Moderately better | 7 | 7
  week 3: A little better | 15 | 27
  week 3: About the same | 36 | 27
  week 3: A little worse | 2 | 1
  week 3: Moderately worse | 1 | 0
  week 3: Much worse | 0 | 2
  week 3: Missing | 2 | 3
  week 4: Much better | 6 | 2
  week 4: Moderately better | 5 | 12
  week 4: A little better | 17 | 20
  week 4: About the same | 35 | 31
  week 4: A little worse | 4 | 2
  week 4: Moderately worse | 0 | 1
  week 4: Much worse | 0 | 1
  week 4: Missing | 3 | 1

28. Secondary Outcome: WPAI-GH Endpoint, Change From Baseline by Timepoint: Absenteeism (%)
Description: The Work Productivity and Activity Impairment questionnaire (WPAI-GH) has 6 questions which address absenteeism, presenteeism (reduced effectiveness while working), overall work productivity loss (absenteeism plus presenteeism), and activity impairment for the 7 days prior to the assessment. WPAI outcomes are presented as impairment percentages (a higher percentage indicating greater impairment and less productivity). Subscale: Absenteeism (work time missed) (%) score, range 0-100.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 4 | -1.24 (22.167) | -5.46 (25.387)
  week 8 | 0.71 (21.429) | -7.75 (28.680)
  week 12 | 6.59 (23.328) | -8.88 (30.513)
  week 16 | 12.43 (28.205) | -7.94 (36.950)
  week 28 | 4.16 (17.279) | -3.59 (40.441)
  week 40 | -1.29 (17.181) | -5.02 (35.641)
  week 52 | 9.02 (23.971) | -10.99 (40.272)

29. Secondary Outcome: WPAI-GH Endpoint, Change From Baseline by Timepoint up to Week 52: Subscale: Presenteeism (Impairment at Work) (%), Range 0-100.
Description: The Work Productivity and Activity Impairment questionnaire (WPAI-GH) has 6 questions which address absenteeism, presenteeism (reduced effectiveness while working), overall work productivity loss (absenteeism plus presenteeism), and activity impairment for the 7 days prior to the assessment. WPAI outcomes are presented as impairment percentages (a higher percentage indicating greater impairment and less productivity). Presenteeism (%) score.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 4 | -7.42 (15.268) | 0.36 (16.439)
  week 8 | -2.58 (15.485) | 6.43 (14.457)
  week 12 | -2.00 (12.247) | 3.20 (20.355)
  week 16 | 2.59 (22.290) | 2.31 (17.043)
  week 28 | -2.41 (19.022) | 3.46 (22.793)
  week 40 | -3.91 (17.252) | 0.43 (10.215)
  week 52 | 4.80 (34.535) | -6.19 (18.568)

30. Secondary Outcome: WPAI-GH Endpoint, Change From Baseline by Timepoint: Work Productivity Loss (%)
Description: The Work Productivity and Activity Impairment questionnaire (WPAI-GH) has 6 questions which address absenteeism, presenteeism (reduced effectiveness while working), overall work productivity loss (absenteeism plus presenteeism), and activity impairment for the 7 days prior to the assessment. WPAI outcomes are presented as impairment percentages (a higher percentage indicating greater impairment and less productivity). Work productivity loss (%) score, range 0-100.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 4 | -7.35 (22.397) | 2.14 (14.775)
  week 8 | -0.53 (23.935) | 6.26 (19.154)
  week 12 | 1.47 (19.235) | 1.24 (24.149)
  week 16 | 8.09 (31.026) | 5.31 (23.864)
  week 28 | 0.05 (25.844) | 6.87 (24.114)
  week 40 | -3.02 (23.350) | 0.67 (14.140)
  week 52 | 5.82 (33.761) | -4.47 (27.803)

31. Secondary Outcome: WPAI-GH Endpoint, Change From Baseline by Timepoint: Activity Impairment (%)
Description: The Work Productivity and Activity Impairment questionnaire (WPAI-GH) has 6 questions which address absenteeism, presenteeism (reduced effectiveness while working), overall work productivity loss (absenteeism plus presenteeism), and activity impairment for the 7 days prior to the assessment. WPAI outcomes are presented as impairment percentages (a higher percentage indicating greater impairment and less productivity). Activity impairment (%) score, range 0-100.
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
score
  week 4 | -3.97 (20.815) | -3.38 (19.745)
  week 8 | -3.53 (21.144) | -4.71 (23.466)
  week 12 | -4.56 (20.620) | -3.97 (20.453)
  week 16 | -3.24 (21.402) | -6.42 (25.268)
  week 28 | -4.41 (22.419) | -6.31 (27.419)
  week 40 | -7.58 (20.234) | -4.46 (20.235)
  week 52 | -3.28 (27.083) | -7.78 (25.492)

32. Secondary Outcome: Absolute Eosinophil Count, Change From Baseline
Description: Absolute eosinophil count, change from baseline by timepoint up to week 52
Time Frame: from baseline to end of DB period, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: cells*10^9/L
Arm/Group | Benralizumab 30 mg | Mepolizumab 300 mg
Number analyzed (Participants) | 70 | 70
cells*10^9/L
  week 1 | 0.15 [0.12 to 0.18] | 0.39 [0.32 to 0.47]
  week 4 | 0.14 [0.12 to 0.17] | 0.30 [0.25 to 0.36]
  week 8 | 0.10 [0.08 to 0.11] | 0.23 [0.20 to 0.28]
  week 12 | 0.11 [0.09 to 0.13] | 0.25 [0.20 to 0.30]
  week 16 | 0.11 [0.09 to 0.13] | 0.24 [0.20 to 0.29]
  week 20 | 0.10 [0.08 to 0.12] | 0.23 [0.19 to 0.28]
  week 24 | 0.14 [0.12 to 0.17] | 0.24 [0.20 to 0.29]
  week 25 | 0.14 [0.11 to 0.17] | 0.23 [0.19 to 0.28]
  week 28 | 0.10 [0.08 to 0.12] | 0.24 [0.20 to 0.29]
  week 32 | 0.12 [0.10 to 0.14] | 0.22 [0.18 to 0.27]
  week 36 | 0.11 [0.09 to 0.14] | 0.26 [0.21 to 0.31]
  week 40 | 0.09 [0.08 to 0.11] | 0.22 [0.18 to 0.27]
  week 44 | 0.10 [0.09 to 0.13] | 0.24 [0.20 to 0.29]
  week 48 | 0.10 [0.08 to 0.13] | 0.24 [0.19 to 0.29]
  week 52 | 0.10 [0.08 to 0.12] | 0.26 [0.21 to 0.32]

ADVERSE EVENTS:
Time Frame: Double-blind Treatment Period: From first dose of study drug until end of Double-blind period, up to 52 weeks. Open-label Extension Period: From the end of the Double-blind period (week 53) to the data cut-off date (10AUG2023), up to 138 weeks.
Description: For analysis of Adverse Events during Double-blind period, Safety Analysis Set is used. Safety Analysis Set: All participants who received at least one dose of Investigational Product (IP). For analysis of Adverse Events during Open-label Extension (OLE) period, OLE Analysis Set is used. OLE Analysis Set: All subjects who entered the OLE part of the study and who received at least 1 dose of IP during the OLE treatment period.
Groups:
- Benra 30 mg - DB: Benralizumab and matching placebo injections delivered subcutaneously every 4 weeks, Double-blind period
- Mepo 300 mg - DB: Mepolizumab and matching placebo injection delivered subcutaneously every 4 weeks, Double-blind period
- Benra 30 mg - OLE: Benralizumab injections delivered subcutaneously every 4 weeks, Open-label extension period (Participants who took Double-blind benralizumab previously)
- Mepo 300 mg Switched to Benra 30 mg - OLE: Benralizumab injections delivered subcutaneously every 4 weeks, Open-label extension period (Participants who took Double-blind mepolizumab previously)
Arm/Group | Benra 30 mg - DB | Mepo 300 mg - DB | Benra 30 mg - OLE | Mepo 300 mg Switched to Benra 30 mg - OLE
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70 | 0/66 | 1/62
Serious Adverse Events (participants affected / at risk) | 4/70 | 9/70 | 10/66 | 13/62
Other Adverse Events (participants affected / at risk) | 46/70 | 56/70 | 43/66 | 46/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg - DB (N=70) | Mepo 300 mg - DB (N=70) | Benra 30 mg - OLE (N=66) | Mepo 300 mg Switched to Benra 30 mg - OLE (N=62)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic infiltration eosinophilic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg - DB (N=70) | Mepo 300 mg - DB (N=70) | Benra 30 mg - OLE (N=66) | Mepo 300 mg Switched to Benra 30 mg - OLE (N=62)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4) | 5 (8) | 7 (9) | 2 (3)
COVID-19 (Infections and infestations) | 14 (14) | 18 (18) | 22 (25) | 27 (30)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (12) | 6 (7) | 11 (19)
Oral candidiasis (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 5 (5) | 8 (9) | 14 (20) | 4 (4)
Sinusitis bacterial (Infections and infestations) | 5 (5) | 3 (4) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4) | 2 (4) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (1) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (6) | 1 (1) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 3 (3) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 8 (8) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 12 (16) | 11 (14) | 1 (1) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 5 (13) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 1 (1) | 5 (5)
Hypertension (Vascular disorders) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (8) | 0 (0) | 0 (0)
Asthenia (General disorders) | 6 (9) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (5) | 6 (7) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 4 (4) | 3 (3) | 7 (10) | 4 (6)
Injection site bruising (General disorders) | 2 (3) | 4 (6) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04157348/Prot_012.pdf
  • Statistical Analysis Plan (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT04157348/SAP_013.pdf